CLINICAL TRIAL: NCT06730659
Title: A Single-Arm, Open-Label, Phase I Study of CHT101 for CD70-Positive Relapsed/Refractory Solid Tumors
Brief Title: A Clinical Study of CHT101 in CD70-Positive Advanced Solid Tumors
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Tianjin Medical University Cancer Institute and Hospital (Other)
Collaborators: Nanjing Calmhome Cell and Gene Engineering Institute Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CHT101SIIT-05
Record Dates: First submitted 2024-12-10; First posted 2024-12-12 (Actual); Last update posted 2024-12-12 (Actual); Status verified 2024-12

CONDITIONS: Relapsed / Refractory Solid Tumor
Keywords: Allogeneic CAR-T; Safety; Efficacy; PK
MeSH Terms: conditions — Recurrence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CHT101 infusion (Experimental): CHT 101 will be dosing by IV.
  Interventions: Biological: CHT101

INTERVENTIONS:
Biological: CHT101 — CHT101: CD 70 UCAR T

SUMMARY:
Evaluate the safety and efficacy of CD70-targeting UCAR-T cells in the treatment of CD70-positive advanced solid tumors.

DETAILED DESCRIPTION:
4 planned dose cohorts will be evaluated during dose escalation phase. The dose expansion will be initiated after SRC (safety review committee) review the avaliable safety, PK and preliminary efficacy data.

ELIGIBILITY:
Inclusion Criteria:

1. Ability to understand and sign a written informed consent documen；
2. At the date of signing ICF, 18 ~70 years old, male or female；
3. Histopathological confirmed advanced or metastatic solid tumors patients who have failed to standard treatment or intolerance with standard treatment；
4. Positive CD70 expression;
5. At least one measurable lesion at baseline per RECIST version 1.1；
6. The expected survival time is more than 12 weeks;
7. ECOG 0-1 points;
8. Adequate organ functions;

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2024-04-19 (Actual); Primary Completion 2027-04-18 (Estimated); Study Completion 2039-04-18 (Estimated)

PRIMARY OUTCOMES:
Safety and Tolerability | 2 years
  Treatment-related adverse events were recorded and assessed according to the National Cancer Institute's Common Terminology Criteria for Adverse Events (CTCAE, Version 5.0)

SECONDARY OUTCOMES:
Objective response rate (ORR) | 28 days
  The proportion of subjects who achieved CR, PR after CAR-T infusion accounted for all treated subjects (Assessed based on RECIST criteria)，the minimum value is 0%，maximum value is 100%, and higher scores mean a better outcome.
Disease control rate (DCR) | 28 days
  The proportion of subjects who achieved CR, PR, SD after CAR-T infusion accounted for all treated subjects (Assessed based on RECIST criteria)，the minimum value is 0%，maximum value is 100%, and higher scores mean a better outcome.
Progress-free survival(PFS) | 2 years
  PFS will be assessed from the first CD70 UCAR-T cell infusion to death from any cause or the first assessment of progression (Assessed based on RECIST criteria)
Overall survival (OS ) | 3 years
  OS will be assessed from the first CD70 UCAR-T cell infusion to death from any cause (Assessed based on RECIST criteria)
pharmacokinetics (PK) | 6 months
  Concentration levels of CD70+ CAR-T cells
Pharmacodynamics (PD) | 6 months
  Concentration levels of CD70 U CAR-T-related serum cytokines, such as IL-2, IL-4, IL-6, IL-10, IFN-γ, TNF-α

CONTACTS AND LOCATIONS:
Locations (1):
- Tianjin Medical University Cancer Institute and Hospital, Tianjin, China

IPD SHARING:
Plan to Share IPD: No